CLINICAL TRIAL: NCT04055701
Title: Relationships Between Preterm Labor and Fetal Thymus Volume in Twin Pregnancies at Second-trimester
Brief Title: Fetal Thymus Volume of Dichorionic Diamniotic Twin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, hidayet şal, assistant doctor, Karadeniz Technical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Fetal Thymus and Preterm labor
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Twin Pregnancy, Antepartum Condition or Complication; Fetal Thymus Volume; Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dichorionic diamniotic twin pregnancy (Other): rutin examination: the assesment of fetal thymus volume at all cases.
  Interventions: Other: assesment of thymus volume

INTERVENTIONS:
Other: assesment of thymus volume — assesment of thymus volume

SUMMARY:
In some studies of fetal thymus volume, fetal stress factors; infection, preterm premature premature rupture of membranes, preeclampsia, preterm delivery risk.

Generally, there is a direct correlation between fetal growth and thymus volume and it was observed that thymus volume decreased in pregnancies accompanied by fetal stress factors.The aim of this study was to measure fetal thymus volume in second trimester twin pregnancies and to investigate whether there is a statistically significant correlation between preterm birth risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Dichorionic di amniotic twin pregnancies between 18 weeks and 23 days 6 days

Exclusion Criteria:

* Single pregnancy,
* first and third trimester pregnant women,
* urinary tract infection, immune system diseases
* fetuses with intrauterine genetic and / or multiple morphological diseases

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
fetal thymus volume | first 6 months
  assesment of volume
fetal thymus volume | last6 months
  assesment of volume
fetal thymus volume | last 6 months
  assesment of volume

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Borgelt JM, Mollers M, Falkenberg MK, Amler S, Klockenbusch W, Schmitz R. Assessment of first-trimester thymus size and correlation with maternal diseases and fetal outcome. Acta Obstet Gynecol Scand. 2016 Feb;95(2):210-6. doi: 10.1111/aogs.12790. Epub 2015 Nov 17. PMID 26445297